CLINICAL TRIAL: NCT06648304
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial to Evaluate the Efficacy and Safety of TTYP01 Tablets in the Treatment of Acute Ischemic Stroke
Brief Title: Evaluate the Efficacy and Safety of TTYP01 Tablets in the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Auzone Biological Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTYP01-III-AIS
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TTYP01 tablets (Experimental): 2 tablets (60 mg) of TTYP01, twice daily, administered 30~60 minutes before breakfast and dinner
  Interventions: Drug: TTYP01 tablets
- Placebo (Simulant TTYP01 Tablets) (Placebo Comparator): 2 tablets (0 mg) of placebo, twice daily, administered 30~60 minutes before breakfast and dinner
  Interventions: Drug: Placebo (Simulant TTYP01 Tablets)

INTERVENTIONS:
Drug: TTYP01 tablets — Administered 30~60 minutes before breakfast and dinner (i.e., fasting state), bid. Subjects are given 2 tablets (60 mg) of investigational drug each time. The first administration should be administered within 1 hour after enrollment. If the subject is randomized in a fed state, the first administration may be administered in a non-fasting state. The interval between the first and second administration should be at least 6 hours, with continuous administration for 28 days (56 administrations).
  Arms: TTYP01 tablets
Drug: Placebo (Simulant TTYP01 Tablets) — Administered 30~60 minutes before breakfast and dinner (i.e., fasting state), bid. Subjects are given 2 tablets (0 mg) of placebo each time. The first administration should be administered within 1 hour after enrollment. If the subject is randomized in a fed state, the first administration may be administered in a non-fasting state. The interval between the first and second administration should be at least 6 hours, with continuous administration for 28 days (56 administrations).
  Arms: Placebo (Simulant TTYP01 Tablets)

SUMMARY:
The study is designed as a multi-center, randomized, double-blind, parallel, placebo-controlled trial to evaluate the efficacy and safety of TTYP01 tablets in the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, parallel, placebo-controlled trial design is used to evaluate the efficacy and safety of TTYP01 tablets in the treatment of patients with acute ischemic stroke.

It is estimated that 618 patients will be enrolled and randomly assigned to the treatment group and the placebo control group in a 1:1 ratio, with 309 patients in each group. Normally, the duration of this study is approximately 90 days. This study will be divided into 2 periods, with a total of five visits: Treatment observation period: D1 ~ D28 (the minimum length of in-hospital observation will be not less than 7 days), including 3 visits (V1- V3); follow-up period: D29 ~ D90, including 2 visits (V4: D60 ± 5 for telephone follow-up; V5: D90 ± 5, returning to hospital for end-of-study visit).

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following inclusion criteria:

1. Patients aged 18 ~ 80 years (both inclusive);
2. Patients diagnosed with acute ischemic stroke according to the 2019AHA/ASA guidelines for ischemic stroke;
3. Patients who do not accept suggestions of thrombolysis or thrombectomy or who do not meet the indications for these treatments;
4. Patients with symptom onset within ≤ 24 hours; for wake-up strokes or when the exact time of symptom onset cannot be determined due to aphasia or disturbance of consciousness, the last time the patient is seen to be normal shall prevail;
5. Patients who are having their first stroke or those who are experiencing a recurrence of stoke after a good recovery (mRS score of 0-1) from their most recent stroke;
6. There are clear signs of neurological deficit: 6≤NIHSS score≤20, and also, the sum of NIHSS score for the 5th upper limb and the 6th lower limb is greater than or equal to 2.
7. Subjects or their guardians are informed about the study, voluntarily agree to the participation, and provide written informed consent.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Patients with any contraindications (such as metal implants like cardiac pacemakers, claustrophobia, etc.) that prevent them from undergoing CT or MRI examinations;
2. Cranial CT or MRI confirmed intracranial hemorrhagic conditions, including but not limited to cerebral hemorrhage, epidural hematoma, subdural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, and traumatic cerebral hemorrhage; or cases of cerebral infarction with post-infarction hemorrhagic transformation. In cases of minor oozing, the investigator will determine eligibility for enrollment;
3. Patients with massive cerebral infarction (low density > 1/3 of the cerebral hemisphere) as indicated by imaging examinations such as CT or MRI;
4. Patients with cerebral infarction accompanied by disturbance of consciousness (NIHSS score Ia > 1 point), posterior circulation infarction, or transient ischemic attack (TIA);
5. Patients with severe mental disorders, depression, or comorbid conditions affecting cognitive function, such as Alzheimer's disease, Parkinson's dementia, or Lewy body dementia, making them unable or unwilling to cooperate with the study;
6. Patients who are scheduled for or have received intravenous thrombolysis, or who require endovascular treatment in the immediate or recent future (within 90 days);
7. Patients with a history of brain malignant tumors or brain parasitic diseases;
8. Patients with a history of severe craniocerebral injury or intracranial infection and an mRS score > 1 prior to this episode;
9. Patients with severe hypertension (systolic blood pressure ≥ 220 mmHg or diastolic blood pressure ≥ 120 mmHg) that is uncontrolled by treatment before the first dose;
10. Patients with blood glucose levels below 2.7 mmol/L without correction or above 22.2 mmol/L at the time of admission;
11. Patients with dysphagia;
12. Patients with a history of rheumatic heart disease or atrial fibrillation; those with a heart rate of less than 40 beats per minute or greater than 120 beats per minute; patients with second or third-degree heart block without a pacemaker or other malignant arrhythmias; and patients who have experienced acute myocardial infarction, cardiac intervention, or heart failure within the past 6 months (classified by the New York Heart Association [NYHA] as III-IV).
13. Patients with other serious systemic or organ diseases that the investigators believe may hinder the evaluation of efficacy or make it unlikely for the patient to complete the expected course of treatment and follow-up (such as malignant tumors with a life expectancy of less than 3 months, etc.).;
14. Patients with severe liver and kidney diseases or abnormal renal and liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] ≥ 3.0 times the upper limit of normal [ULN]; serum creatinine [Cr] > 2.0 times the ULN);
15. Patients with a bleeding tendency, including platelet count (PLT) less than 75.0×10^9/L, or severe bleeding within the 3 months prior to the onset of the disease.
16. Patients with contraindications to antiplatelet therapy or statin therapy;
17. Patients with allergic constitution, hypersensitivity to Edaravone or its excipients;
18. Patients with suspected or confirmed history of alcohol or drug abuse;
19. Patients who are pregnant, lactating or have a recent pregnancy plan and are unwilling to use contraception;
20. Patients who have participated in other clinical trials within 3 months or are participating in other clinical studies prior to this study;
21. Patients who are deemed unsuitable by the investigator for participation in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with mRS score ≤1 on Day 90 of treatment. | 90 days after treatment initiation
  The mRS (modified Rankin Scale) is a scoring system used to assess the ability of post-stroke patients in their daily lives. It assesses the degree of functional impairment of patients after stroke through a standardized questionnaire, and is one of the most widely used tools for assessing the sequelae of stroke internationally. The MRS scores range from 0 to 5, with higher scores indicating more severe disability in patients.

SECONDARY OUTCOMES:
mRS score on Day 90 of treatment | 90 days after treatment initiation
  The mRS (modified Rankin Scale) is a scoring system used to assess the ability of post-stroke patients in their daily lives. It assesses the degree of functional impairment of patients after stroke through a standardized questionnaire, and is one of the most widely used tools for assessing the sequelae of stroke internationally. The MRS scores range from 0 to 5, with higher scores indicating more severe disability in patients.
Proportion of subjects with mRS score ≤2 on D90 of treatment | 90 days after treatment initiation
  The mRS (modified Rankin Scale) is a scoring system used to assess the ability of post-stroke patients in their daily lives. It assesses the degree of functional impairment of patients after stroke through a standardized questionnaire, and is one of the most widely used tools for assessing the sequelae of stroke internationally. The MRS scores range from 0 to 5, with higher scores indicating more severe disability in patients.
Change from baseline in mRS score on D7, D28, D60 and D90 of treatment | Baseline and 7, 28, 60, 90 days after treatment initiation
  The mRS (modified Rankin Scale) is a scoring system used to assess the ability of post-stroke patients in their daily lives. It assesses the degree of functional impairment of patients after stroke through a standardized questionnaire, and is one of the most widely used tools for assessing the sequelae of stroke internationally. The MRS scores range from 0 to 5, with higher scores indicating more severe disability in patients.
Change in NIHSS score from baseline on D7, D28 and D90 of treatment | Baseline and 7, 28, 90 days after treatment initiation
  The NIHSS (National Institutes of Health Stroke Scale) is a standardized neurological examination tool used to assess neurological deficits in stroke patients. The scale consists of 15 tests and the total score is the sum of the individual scores ranges from 0 to 42, with lower scores indicating a better state of the patient.
Proportion of patients with NIHSS score improvement ≥ 4 points on D7, D28, and D90 of treatment | 7, 28 and 90 days after treatment initiation
  The NIHSS (National Institutes of Health Stroke Scale) is a standardized neurological examination tool used to assess neurological deficits in stroke patients. The scale consists of 15 tests and the total score is the sum of the individual scores ranges from 0 to 42, with lower scores indicating a better state of the patient.
Proportion of subjects with NIHSS score of 0-1 on D7, D28 and D90 of treatment | 7, 28 and 90 days after treatment initiation
  The NIHSS (National Institutes of Health Stroke Scale) is a standardized neurological examination tool used to assess neurological deficits in stroke patients. The scale consists of 15 tests and the total score is the sum of the individual scores ranges from 0 to 42, with lower scores indicating a better state of the patient.
Change in BI score from baseline on D7, D28 and D90 of treatment | Baseline and 7, 28, 90 days after treatment initiation
  The BI (Barthel Index) is used to assess the patient's ability to perform activities of daily living and can be used to evaluate the patient's functional recovery before and after treatment, and it is one of the most widely used and researched methods of basic assessment of activities of daily living in clinical practice, with credible results. It is mainly based on the patient's actual daily performance and is not judged by the ability the patient may have. The BI scores range from 0 to 100, with higher scores indicating a better state of the patient.
Proportion of subjects with BI score ≥ 95 points on D7, D28 and D90 of treatment | 7, 28 and 90 days after treatment initiation
  The BI (Barthel Index) is used to assess the patient's ability to perform activities of daily living and can be used to evaluate the patient's functional recovery before and after treatment, and it is one of the most widely used and researched methods of basic assessment of activities of daily living in clinical practice, with credible results. It is mainly based on the patient's actual daily performance and is not judged by the ability the patient may have. The BI scores range from 0 to 100, with higher scores indicating a better state of the patient.
MoCA score and comparison on D7, D28 and D90 of treatment | 7, 28 and 90 days after treatment initiation
  The MoCA (Montreal Cognitive Assessment) Scale is a rating tool used to provide rapid screening for cognitive dysfunction. It includes 11 screening items in 8 cognitive domains: attention and concentration, executive function, memory, language, visual structural skills, abstract thinking, calculation and orientation. The total score is 30, with ≥26 being normal; the lower the score, the more severe the cognitive impairment.
HDRS score and comparison on D7, D28 and D90 of treatment | 7, 28 and 90 days after treatment initiation
  The HDRS (Hamilton Depression Scale) was developed by Hamilton in 1960 and is the most commonly used scale for assessing depressive states in clinical settings. There are three versions of this scale: 17-item, 21-item and 24-item. The 21-item version was used for this Clinical Study, with a score range from 0 to 64. A score greater than 30 is severe depression, greater than 20 is moderate depression, and greater than 17 is mild depression.
Proportion of subjects with recurrent stroke within 90 days of treatment | within 90 days of treatment
Changes in cranial MRI findings (infarct volume) relative to baseline | Baseline and 5, 28 days after treatment initiation
  Infarct volume will report in mm^3
Changes in cranial MRI findings (infarct area) relative to baseline | Baseline and 5, 28 days after treatment initiation
  Infarct area will report in mm^2

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Jiang Wang, MD & PhD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China

DOCUMENTS (3):
  • Study Protocol: V2.0 (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT06648304/Prot_000.pdf
  • Study Protocol: V1.0 (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT06648304/Prot_001.pdf
  • Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT06648304/SAP_002.pdf